CLINICAL TRIAL: NCT05165758
Title: Comparison of the Quality of Life and the Level of Precarity of a Diabetic Population With and Without Foot Ulcer in Martinique
Acronym: QVP-Dia
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 21_RIPH3-04
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Diabetes; Diabetes Mellitus; Foot Ulcer, Diabetic; Diabetes Complications
Keywords: Diabete; Diabete complications; Diabetic foot ulcer; socio-economic disparities
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic subjects without foot ulcer: 27 diabetic subjects without foot ulcer will answer to the SF-36 score (mental health items) and to a french precarit index (EPICES:Evaluation de la précarité et des inégalités de santé dans les Centres d'examens de santé)
  Interventions: Other: Self-assessment questionnaires
- Diabetic subjects with foot ulcer: 54 diabetic subjects presenting foot ulcer will answer to the SF-36 score (mental health items) and to a french precarit index (EPICES:Evaluation de la précarité et des inégalités de santé dans les Centres d'examens de santé)
  Interventions: Other: Self-assessment questionnaires

INTERVENTIONS:
Other: Self-assessment questionnaires — Subjects will pass the SF-36 score (mental health items) and the EPICES index

SUMMARY:
The aim of this study is to compare quality of life of diabetics with and without foot ulcer. Investigators will compare their quality of life based on the mental health impact of foot ulcer.

DETAILED DESCRIPTION:
Diabetes is one of the most frequent pathologies in Martinique (French West Indies) in terms of prevalence, as are its complications. The diabetic foot ulcer is a real public health problem considering its impact on the island.

It has already been shown that diabetic patients have a lower quality of life than the overall population. It is now time to compare the quality of life of diabetics with and without foot ulcer in Martinique.

Such a complication has a social impact that should not be overlooked in primary, secondary and tertiary prevention.

ELIGIBILITY:
Inclusion Criteria:

* People of 18 years old and over,
* Diabetics living in Martinique,
* Patient having been informed of the research,
* Patient agreeing to participate in the study.

Exclusion Criteria:

* Minor patient,
* Hospitalized patients during inclusion phase,
* Patients with confusional syndrome,
* Patient presenting a cognitive state making it difficult to complete the questionnaire,
* Patient under legal protection, under guardianship or under curatorship,
* Patient who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic subjects
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Compare the levels of quality of life in diabetic subjects with and without foot ulcer | 6 months
  The primary endpoint will be the score on the mental health dimension of the SF-36 score

SECONDARY OUTCOMES:
Compare the levels of precarity in diabetic subjects with and without foot ulcer | 6 months
  To evaluate the level of precarity, the EPICES score will be calculated for both type of subjects.
Compare the levels of quality of life according to the levels of HbA1c, in diabetic subjects with and without foot ulcer | 6 months
  To evaluate the level of quality of life according to HbA1c, the score of the mental health dimension of the SF-36 questionnaire will be calculated for both type of subjects.
Compare the quality of life levels according to the duration of diabetes, in diabetic subjects with and without foot ulcer | 6 months
  To evaluate the level of quality of life according to the duration of diabetes, the score of the mental health dimension of the SF-36 questionnaire will be calculated for both type of subjects.
Compare the quality of life levels according to the type of antidiabetic treatment, in diabetic subjects with and without foot ulcer | 6 months
  To evaluate the level of quality of life according to the antidiabetic treatment, the score of the mental health dimension of the SF-36 questionnaire will be calculated for both type of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel BOURGADE, MD, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, Martinique, France

IPD SHARING:
Plan to Share IPD: No